CLINICAL TRIAL: NCT04827056
Title: Effect of Sublingual Formulation of Dexmedetomidine HCl (BXCL501) on Ethanol in Heavy Drinkers With PTSD - Alcohol Interaction Study
Brief Title: Effect of Sublingual Formulation of Dexmedetomidine HCl (BXCL501) - Alcohol Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacotherapies for Alcohol and Substance Use Disorders Alliance (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency); RTI International (Other); VA Connecticut Healthcare System (U.S. Federal Agency); BioXcel Therapeutics Inc (Industry); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: AS170014-A7; W81XWH1820044 (Other Grant/Funding Number: Department of Defense Congressionally Directed Medical Research Program)
Record Dates: First submitted 2021-03-17; First posted 2021-04-01 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Alcohol Use Disorder (AUD); Post Traumatic Stress Disorder (PTSD)
Keywords: Alcohol Used Disorder (AUD); Post Traumatic Stress Disorder; Alcohol Use; Heavy Drinkers; Dexmedetomidine HCl (BXCL501)
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic; Alcohol Drinking | interventions — Dexmedetomidine; Organization and Administration; Ethanol

STUDY DESIGN:
Intervention Model Description: All participants will be randomized to receive BXCL501 40µg, 80µg or placebo in a modified crossover randomization scheme in which all participants will receive each possible study drug assignment but must receive 40µg before receiving the higher dose (80µg).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Apart from the Research Pharmacists, all others engaged with this study (participants and study team) will be masked to the drug sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine (DEX) for sublingual (SL) administration (BXCL501) - 40µg (Experimental): BXCL501 is a thin film formulation of dexmedetomidine (DEX) for sublingual (SL) administration. The product is a small, solid-dose film formulation, approximately 286 mm2 in area and 0.7 mm thick, designed to solubilize in the SL space within 1-3 minutes. At the time of dosing, subjects will be verbally instructed on how to take the investigational product sublingually, and that they should retain the investigational product in the sublingual cavity until dissolved.
  Interventions: Drug: Placebo; Drug: Dexmedetomidine (DEX) for sublingual (SL) administration (BXCL501) - 40µg; Drug: Dexmedetomidine (DEX) for sublingual (SL) administration (BXCL501) - 80µg; Procedure: Ethanol Infusion; Behavioral: PTSD Reactivity Condition; Behavioral: Alcohol Cue Reactivity
- Dexmedetomidine (DEX) for sublingual (SL) administration (BXCL501) - 80µg (Experimental): BXCL501 is a thin film formulation of dexmedetomidine (DEX) for sublingual (SL) administration. The product is a small, solid-dose film formulation, approximately 286 mm2 in area and 0.7 mm thick, designed to solubilize in the SL space within 1-3 minutes. At the time of dosing, subjects will be verbally instructed on how to take the investigational product sublingually, and that they should retain the investigational product in the sublingual cavity until dissolved.
  Interventions: Drug: Placebo; Drug: Dexmedetomidine (DEX) for sublingual (SL) administration (BXCL501) - 40µg; Drug: Dexmedetomidine (DEX) for sublingual (SL) administration (BXCL501) - 80µg; Procedure: Ethanol Infusion; Behavioral: PTSD Reactivity Condition; Behavioral: Alcohol Cue Reactivity
- Placebo (Placebo Comparator): Placebo and study drug will look exactly the same in order to maintain the double-blind; study drug and placebo are administered exactly the same.
  Interventions: Drug: Placebo; Drug: Dexmedetomidine (DEX) for sublingual (SL) administration (BXCL501) - 40µg; Drug: Dexmedetomidine (DEX) for sublingual (SL) administration (BXCL501) - 80µg; Procedure: Ethanol Infusion; Behavioral: PTSD Reactivity Condition; Behavioral: Alcohol Cue Reactivity

INTERVENTIONS:
Drug: Placebo — Placebo will be administered orally, as individual films in the SL space.
Drug: Dexmedetomidine (DEX) for sublingual (SL) administration (BXCL501) - 40µg — BXCL 501 40µg will be administered orally, as individual films in the SL space.
  Other Names: BXCL501 40µg
Drug: Dexmedetomidine (DEX) for sublingual (SL) administration (BXCL501) - 80µg — BXCL 501 80µg will be administered orally, as individual films in the SL space.
  Other Names: BXCL501 80µg
Procedure: Ethanol Infusion — Study team will be using a modified alcohol-IV clamp procedure developed and standardized by Subramanian and colleagues (Subramanian, Heil et al. 2002). The infusion will be performed using a 6% ethanol solution in 0.9% saline. The computer assisted administration program automatically calculates and corrects the infusion rate based on real-time BrAC data entry by staff, based on the pharmacokinetic profile of each subject (targeting a breath alcohol concentration (BrAC) of 100 mg%).
Behavioral: PTSD Reactivity Condition — Participants will be exposed to two conditions in random order: PTSD cues and neutral cues. The cues will consist of a 5 minute presentation of the stimulus (trauma or neutral) followed by immediate evaluation of craving and anxiety. There will be a relaxation procedure between each condition. The imagery scripts are developed based on the scene construction questionnaire developed by Lang et al (Lang, Kozak et al. 1980, Lang, Levin et al. 1983) using a standardized format designed by Sinha (Sinha 2001).
Behavioral: Alcohol Cue Reactivity — Participants will be exposed to two conditions: a neutral cue (water) followed by an alcohol cue. Individuals will be instructed that they may smell and handle the beverage, but they cannot consume the beverage. Following the presentation, the research assistant takes the beverage and leaves the room, while the subject completes the anxiety and alcohol craving assessments.

SUMMARY:
The overall objective of the proposed study is to determine if Dexmedetomidine HCl (BXCL501) is safe for treatment of alcohol use disorder (AUD) with comorbid posttraumatic stress disorder (PTSD) and also shows potential signals of efficacy thereby supporting the conduct of later phase clinical trials. Safety endpoints will be compared following an alcohol challenge without and concurrent with BXCL501 treatment.

DETAILED DESCRIPTION:
BXCL501 is a sublingual film containing dexmedetomidine. Dexmedetomidine is an alpha-2 adrenergic receptor agonist and has higher intrinsic activity and is more potent in vitro than either clonidine or lofexidine. The drug has a high free brain to free plasma ratio after dosing in rats that persists after plasma concentrations are cleared. Dexmedetomidine does not depress respiratory function. It is not predicted to have abuse potential. BXCL501 will bypass 1st pass metabolism and produce fewer problems in participants with compromised liver function.

This laboratory study is a phase 1, double-blind, placebo-controlled, within subjects study. This study will consist of 3 laboratory test sessions following pretreatment with BXCL501/placebo for 10 heavy drinker participants with comorbid PTSD. Participants (n=10) will participate in a laboratory study with 3 test days (minimum of 2 days, but no longer than 2 weeks between each test session); for each test day they will be assigned to receive sublingual BXCL501 40µg, 80µg and placebo in a randomized fashion. Test sessions will be conducted to evaluate stress (PTSD) reactivity and alcohol cue reactivity. Participants will also receive IV ethanol administered via "clamp methodology" to assess for the effects of BXCL501 in combination with ethanol.

Since this is the first time BXCL501 is being tested in combination with alcohol administration, the study team will be using a modified randomization where participants will not receive the 80µg dose until they have received the 40µg dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, Veterans and non-Veterans, ages 21 to 65;
2. Able to read and write in English and sign the informed consent;
3. Willing to comply with all study procedures and be available for the duration of the study;
4. ECG that demonstrates no clinically significant conduction issues or arrhythmias;
5. Have no clinically significant contraindications, in the judgement of the PI/study physician, for study participation (based on self-reported medical history and brief physical examination);
6. Have a current diagnosis of Alcohol use disorder (AUD) (mild, moderate, or severe) as determined by MINI-5
7. Have a traumatic event in their lifetime that meets Criterion A for PTSD;
8. Must have > 1 heavy drinking episodes (>4 standard drink units (SDU) for men; >3 SDU for women) in the last 30 days (assessed by the Timeline Follow Back (TLFB)).
9. Not be treatment seeking for AUD
10. Females of childbearing potential (not surgically sterilized (tubal ligation/hysterectomy) or not post-menopausal (no menstrual period for > 6 months) must be willing to use a medically acceptable and effective birth control method for 3 months before the study and while participating in the study. Medically acceptable methods of contraception that may be used by the participant include abstinence, birth control pills or patches, birth control implants, diaphragm, intrauterine device (IUD), or condoms.

Exclusion Criteria:

1. Current bipolar disorder or psychotic disorders as determined by MINI-5;
2. Current diagnosis of a substance use disorder (other than alcohol, nicotine, or marijuana) as determined by MINI-5;
3. Females who are pregnant, nursing, or planning to become pregnant during study participation;
4. Current physiological alcohol dependence requiring a higher level of care (e.g. detox) as determined by study physician conducting physical examination and CIWA score. Tolerance to alcohol will be allowed.
5. Recent history of complicated alcohol withdrawal, alcohol withdrawal seizures, or delirium tremens (DTs);
6. Score > 4 on Clinical Institute Withdrawal Assessment for Alcohol Scale (CIWA-Ar) at randomization;
7. History of major medical illnesses including liver disease, heart disease, chronic pain or other medical conditions that the physician investigator deems contraindicated for the participant to be in the study;
8. Clinically significant history of cardiac disease including (a) chronic hypertension (even if adequately controlled by antihypertensive medications); (b) history of syncope or other syncopal attacks; (c) current evidence of orthostatic hypotension (defined as a decrease in systolic BP of 20 mm Hg or decrease in diastolic BP of 10mm Hg within 3 minutes); (d) resting heart rate of <60 beats per minute; (e) systolic blood pressure <110mmHg or diastolic BP <70mmHg; or (f) participants with a QTC interval >440msec (males) or >460msec (females).
9. Clinically significant medical conditions including hepatic ascites (bilirubin >10% above the upper limit of normal [ULN] or liver function tests [LFT] >3 × ULN);
10. Renal impairment as measured by BUN/Creatinine;
11. Currently taking the following medications: a) medications for alcoholism (e.g. naltrexone, disulfiram, topiramate, acamprosate); b) psychotropic medications that promote sedation including sedative/hypnotics, barbiturates, antihistamines, sedative antidepressants (e.g. doxepin, mirtazapine, trazodone), and triptans (e.g., sumatriptan); c) antihypertensive medications; d) alpha-2-adrenergic agonists (clonidine, guanfacine, lofexidine); or adrenergic agents prescribed for other reasons are excluded (prazosin). (Permitted Concomitant Medications: The concomitant medications allowed in the study include non-sedative antidepressants used to treat PTSD);
12. History of allergic reactions to dexmedetomidine or known allergy to dexmedetomidine;
13. Participation in a clinical trial of a pharmacological agent within 30 days prior to screening;
14. Any finding that, in the view of the principal investigator, would compromise the subject's ability to fulfill the study visit schedule or requirements

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Change in anxiety, as measured by blood pressure (systolic and diastolic), by treatment group during stress reactivity conditions. | On each Test Day (1-3), from baseline (prior to stress condition) to the end of the PTSD stress reactivity conditions
  Anxiety is measured via blood pressure (systolic and diastolic). Participants will undergo stress (PTSD) reactivity conditions (both neutral and trauma) on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in blood pressure is computed as the difference in measurements taken across the PTSD Reactivity Conditions to the measurement collected immediately prior to the stress condition.
Change in anxiety, as measured by heart rate, by treatment group during stress reactivity conditions. | On each Test Day (1-3), from baseline (prior to stress condition) to the end of the PTSD stress reactivity conditions .
  Anxiety is measured via heart rate. Participants will undergo stress (PTSD) reactivity conditions (both neutral and trauma) on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in heart rate is computed as the difference in measurements taken across the PTSD Reactivity Conditions to the measurement collected immediately prior to the stress condition.
Change in anxiety, as measured by the State Trait Anxiety Inventory (STAI-6), by treatment group during stress reactivity conditions. | On each Test Day (1-3), from baseline (prior to stress condition) to the end of the PTSD stress reactivity conditions.
  Anxiety is measured via the State Trait Anxiety Inventory (STAI-6). Participants will undergo stress (PTSD) reactivity conditions (both neutral and trauma) on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in STAI-6 score is computed as the difference in measurements taken across the PTSD Reactivity Conditions to the measurement collected immediately prior to the stress condition.
Change in alcohol craving, as measured by the Yale Craving Scale (YCS), by treatment group during stress reactivity conditions. | On each Test Day (1-3), from baseline (prior to stress condition) to the end of the PTSD stress reactivity conditions.
  Alcohol craving is measured via the Yale Craving Scale (score range is 0 to 112, with 0 meaning "no sensation" and 112 meaning "strongest imaginable sensation of any kind"). Participants will undergo stress (PTSD) reactivity conditions (both neutral and trauma) on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in YCS is computed as the difference in measurements taken across the PTSD Reactivity Conditions to the measurement collected immediately prior to the stress condition.
Change in mood disturbance, as measured by Drugs Effects Questionnaire (DEQ), by treatment group during stress reactivity conditions. | On each Test Day (1-3), from baseline (prior to stress condition) to the end of the PTSD stress reactivity conditions.
  Mood disturbance is measured via the Drugs Effects Questionnaire (DEQ). Participants will undergo stress (PTSD) reactivity conditions (both neutral and trauma) on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in DEQ is computed as the difference in measurements taken across the PTSD Reactivity Conditions to the measurement collected immediately prior to the stress condition.
Change in mood disturbance, as measured by Visual Analog Scale (VAS), by treatment group during stress reactivity conditions. | On each Test Day (1-3), from baseline (prior to stress condition) to the end of the PTSD stress reactivity conditions.
  Mood disturbance is measured via the Visual Analog Scale (score range is 0 to 100, with 0 having no specific mood disturbance and 100 having extreme specific mood disturbance). Participants will undergo stress (PTSD) reactivity conditions (both neutral and trauma) on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in VAS is computed as the difference in measurements taken across the PTSD Reactivity Conditions to the measurement collected immediately prior to the stress condition.
Change in anxiety, as measured by blood pressure (systolic and diastolic), by treatment group during alcohol cue induced craving. | On each Test Day (1-3), from baseline (prior to alcohol reactivity conditions) to assessments conducted immediately after the alcohol reactivity conditions.
  Anxiety is measured via blood pressure (systolic and diastolic). Participants will undergo an alcohol cue reactivity condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in blood pressure is computed as the difference in measurements taken across the alcohol reactivity conditions to the measurement collected immediately prior to the alcohol reactivity condition.
Change in anxiety, as measured by heart rate, by treatment group during alcohol cue induced craving. | On each Test Day (1-3), from baseline (prior to alcohol reactivity conditions) to assessments conducted immediately after the alcohol reactivity conditions.
  Anxiety is measured via heart rate. Participants will undergo an alcohol cue reactivity condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in heart rate is computed as the difference in measurements taken across the alcohol reactivity conditions to the measurement collected immediately prior to the alcohol reactivity condition.
Change in anxiety, as measured by the State Trait Anxiety Inventory (STAI-6), by treatment group during alcohol cue induced craving. | On each Test Day (1-3), from baseline (prior to alcohol reactivity conditions) to assessments conducted immediately after the alcohol reactivity conditions.
  Anxiety is measured via the State Trait Anxiety Inventory (STAI-6). Participants will undergo an alcohol cue reactivity condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in STAI-6 score is computed as the difference in measurements taken across the alcohol reactivity conditions to the measurement collected immediately prior to the alcohol reactivity conditions.
Change in alcohol craving, as measured by the Yale Craving Scale (YCS), by treatment group during alcohol cue induced craving. | On each Test Day (1-3), from baseline (prior to alcohol reactivity conditions) to assessments conducted immediately after the alcohol reactivity conditions.
  Alcohol craving is measured via the Yale Craving Scale (score range is 0 to 112, with 0 meaning "no sensation" and 112 meaning "strongest imaginable sensation of any kind"). Participants will undergo an alcohol cue reactivity condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in YCS is computed as the difference in measurements taken across the alcohol reactivity conditions to the measurement collected immediately prior to the alcohol reactivity conditions
Change in mood disturbance, as measured by Drugs Effects Questionnaire (DEQ), by treatment group during alcohol cue induced craving. | On each Test Day (1-3), from baseline (prior to alcohol reactivity conditions) to assessments conducted immediately after the alcohol reactivity conditions.
  Mood disturbance is measured via the Drugs Effects Questionnaire (DEQ). Participants will undergo an alcohol cue reactivity condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in DEQ is computed as the difference in measurements taken across the alcohol cue reactivity condition to the measurement collected immediately prior to the alcohol cue reactivity condition.
Change in mood disturbance, as measured by Visual Analog Scale (VAS), by treatment group during alcohol cue induced craving. | On each Test Day (1-3), from baseline (prior to alcohol reactivity conditions) to assessments conducted immediately after the alcohol reactivity conditions.
  Mood disturbance is measured via the Visual Analog Scale (score range is 0 to 100, with 0 having no specific mood disturbance and 100 having extreme specific mood disturbance). Participants will undergo an alcohol cue reactivity condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in VAS is computed as the difference in measurements taken across the alcohol cue reactivity condition to the measurement collected immediately prior to the alcohol cue reactivity condition.
Evaluate whether pretreatment with BXCL501 alters subjective effects, as measured by the Biphasic Alcohol Effects Scale (BAES), in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to alcohol infusion start) to assessments conducted immediately after the alcohol infusion.
  The BAES is a 14-item self-report adjective rating scale that will serve to measure stimulant and sedative effects of alcohol. The Stimulation subscale score range is 0 to 70, with higher scores indicating greater stimulation. The Sedation subscale score range is 0 to 70, with higher scores indicating greater sedation. Participants will undergo alcohol infusion condition on laboratory test days 1, 2, and 3 (receiving either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), change in BAES score is computed as the difference in measurements taken across the alcohol infusion to the measurement collected immediately prior to the alcohol infusion. Differences in the change in BAES score will be compared across all three treatment arms.
Evaluate whether pretreatment with BXCL501 alters subjective effects, as measured by the Number of Drinks Scale (NDS), in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to alcohol infusion start) to assessments conducted immediately after the alcohol infusion.
  Self-rated alcohol intoxication is measured by the Number of Drinks Scale (NDS). The NDS assess how many drinks the subject feels he/she has consumed at a specific timepoint (the higher the number the greater the alcohol intoxication). Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in NDS score is computed as the difference in measurements taken across the alcohol infusion to the measurement collected immediately prior to the alcohol infusion. Differences in the change in NDS score will be compared across all three treatment arms.
Evaluate whether pretreatment with BXCL501 alters subjective effects, as measured by the State Trait Anxiety Inventory (STAI-6), in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to alcohol infusion start) to assessments conducted immediately after the alcohol infusion.
  The STAI-6 is a 6-item measure designed to assess trait and state aspects of anxiety. Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in STAI-6 score is computed as the difference in measurements taken across the alcohol infusion to the measurement collected immediately prior to the alcohol infusion. Differences in the change in STAI-6 score will be compared across all three treatment arms.
Evaluate whether pretreatment with BXCL501 alters subjective effects, as measured by the Drug Effects Questionnaire (DEQ), in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to alcohol infusion start) to assessments conducted immediately after the alcohol infusion.
  The DEQ is a 5-item self-report measure used to assess the two key aspects of the subjective experience of substance effects: (1) the strength of substance effects and (2) the desirability of substance effects. Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in DEQ score is computed as the difference in measurements taken across the alcohol infusion to the measurement collected immediately prior to the alcohol infusion. Differences in the change in DEQ score will be compared across all three treatment arms.
Evaluate whether pretreatment with BXCL501 alters subjective effects, as measured by the Yale Craving Scale (YCS), in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to alcohol infusion start) to assessments conducted immediately after the alcohol infusion.
  Alcohol craving is measured via the Yale Craving Scale (score range is 0 to 112, with 0 meaning "no sensation" and 112 meaning "strongest imaginable sensation of any kind"). Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in YCS score is computed as the difference in measurements taken across the alcohol infusion to the measurement collected immediately prior to the alcohol infusion. Differences in the change in YCS score will be compared across all three treatment arms.
Evaluate whether pretreatment with BXCL501 alters subjective effects, as measured by the Visual Analog Scale (VAS), in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to alcohol infusion start) to assessments conducted immediately after the alcohol infusion.
  Mood disturbance is measured via the Visual Analog Scale (score range is 0 to 100, with 0 having no specific mood disturbance and 100 having extreme specific mood disturbance). Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in VAS score is computed as the difference in measurements taken across the alcohol infusion to the measurement collected immediately prior to the alcohol infusion. Differences in the change in VAS score will be compared across all three treatment arms.
Evaluate whether pretreatment with BXCL501 alters motor impairment, as measured by the Grooved Pegboard (GPB), in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to drug administration) to assessments conducted immediately after the alcohol infusion.
  The GPB is a manipulative dexterity test, consisting of a board with randomly positioned slots in which subjects insert pegs. It is an eye-to-hand coordination test that has been used in research studies to measure motor skills. Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in GPB score is computed as the difference in measurements taken across the alcohol infusion to the measurement collected immediately prior to drug administration. Differences in the change in GPB score will be compared across all three treatment arms.
Evaluate whether pretreatment with BXCL501 alters cognitive functioning, as measured by the Rapid Information Processing Task (RVIP), in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to drug administration) to the RVIP assessment conducted immediately after the targeted BAL is reached during the alcohol infusion.
  The RVIP is a widely used task to assess sustained attention, with a working memory component. These cognitive functions are sensitive to acute alcohol administration. Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in RVIP score is computed as the difference in the RVIP measurement taken once the targeted BAL is achieved during the alcohol infusion to the measurement collected immediately prior to drug administration.
Evaluate whether pretreatment with BXCL501 alters cognitive functioning, as measured by the Hopkins Verbal Learning Test-Revised (HVLT-R), in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to drug administration) to the HVLT-R assessment conducted immediately after the targeted BAL is reached during the alcohol infusion.
  The HVLT-R is a word list learning test of verbal memory and is sensitive to the acute effects of alcohol. Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in HVLT-R score is computed as the difference in the HVLT-R measurement taken once the targeted BAL is achieved during the alcohol infusion to the measurement collected immediately prior to drug administration.
Evaluate whether pretreatment with BXCL501 alters cognitive functioning, as measured by the Go No-Go Task, in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to drug administration) to the Go No-Go assessment conducted immediately after the targeted BAL is reached during the alcohol infusion.
  The Go No-Go task will assess the ability to withhold responses to an infrequently occurring target (No-Go trials). Alcohol has been shown to impair responses to Go No-Go task. Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in Go No-Go score is computed as the difference in the Go No-Go measurement taken once the targeted BAL is achieved during the alcohol infusion to the measurement collected immediately prior to drug administration.
Evaluate whether pretreatment with BXCL501 increases side effects, as measured by blood pressure (systolic and diastolic), in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to alcohol infusion) to the blood pressure measurement taken after completion of the alcohol infusion.
  Potential side-effects of BXCL501 in the presence of alcohol will be measured via blood pressure. Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in blood pressure is computed as the difference in measurements taken across the alcohol infusion to the measurement collected immediately prior to the alcohol infusion.
Evaluate whether pretreatment with BXCL501 increases side effects, as measured by heart rate, in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to alcohol infusion) to the heart rate measurement taken after completion of the alcohol infusion.
  Potential side-effects of BXCL501 in the presence of alcohol will be measured via heart rate. Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in heart rate is computed as the difference in measurements taken across the alcohol infusion to the measurement collected immediately prior to the alcohol infusion.
Evaluate whether pretreatment with BXCL501 increases side effects, as measured by the Richmond Agitation Sedation Scale (RASS), in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to alcohol infusion) to the RASS measurement taken after completion of the alcohol infusion.
  Potential side-effects of BXCL501 in the presence of alcohol will be measured via the RASS, which is assessed by clinic staff to measure participant's level of sedation. The score range is +4 (combative) to -5 (unarousable), thus lower scores indicate greater sedation. Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in RASS score is computed as the difference in measurements taken across the alcohol infusion to the measurement collected immediately prior to the alcohol infusion.
Evaluate whether pretreatment with BXCL501 increases side effects, as measured by the Agitation-Calmness Evaluation Scale (ACES), in the presence of ethanol. | On each Test Day (1-3), from baseline (prior to alcohol infusion) to the ACES measurement taken after completion of the alcohol infusion.
  Potential side-effects of BXCL501 in the presence of alcohol will be measured via the ACES, which is assessed by clinic staff to measure participants' level of sedation. The score range is 1 (marked agitation) to 9 (unarousable), thus higher scores indicate greater sedation. Participants will undergo an alcohol infusion condition on laboratory test days 1, 2, and 3 (where participant receives either BXCL501 40µg, 80µg, or placebo in a randomized fashion each day). For each test day (1-3), the change in ACES score is computed as the difference in measurements taken across the alcohol infusion to the measurement collected immediately prior to the alcohol infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Ismene Petrakis, MD, Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No